CLINICAL TRIAL: NCT05459688
Title: An Open-Label Extension Study of Patients Previously Enrolled in Study CIN-107-124 to Evaluate the Long-Term Safety and Effectiveness of CIN-107
Brief Title: Open-Label Extension Study of Patients Previously Enrolled in Study CIN-107-124
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIN-107-130; D6971C00001 (Other: AstraZeneca)
Record Dates: First submitted 2022-06-17; First posted 2022-07-15 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Eligible patients from Study CIN-107-124 who elect to participate in this study will continue treatment with 2 mg CIN-107 tablets QD after enrollment, starting at Visit 1 and concluding at EOT (Visit 7)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental 2 mg CIN-107 tablets QD (Experimental): Treatment with 2 mg CIN-107 tablets, by mouth, once per day. Starting at Visit 1 and concluding at EOT (Visit 7).
  Interventions: Drug: CIN-107

INTERVENTIONS:
Drug: CIN-107 — 2 mg of CIN-107, once a day for 52 weeks

SUMMARY:
This is a Phase 2, multicenter, open-label extension (OLE) study to evaluate the long-term safety, tolerability, and effectiveness of CIN-107 for up to 52 weeks in patients with HTN who have completed Part 1 or Part 2 of Study CIN-107-124. The study will be conducted at clinical sites that have participated in the double-blind, Phase 2 Study CIN-107-124.

ELIGIBILITY:
Inclusion Criteria:

1. Have completed Part 1 or Part 2 of Study CIN-107-124;
2. Have had acceptable safety and tolerability during Study CIN-107-124 as determined by the Investigator or Medical Monitor;
3. Have demonstrated ≥70% and ≤120% adherence to their single background antihypertensive agent and the CIN-107 placebo during Study CIN-107-124;
4. Agree to comply with the contraception and reproduction restrictions of the study as follows:

   * Male patients must agree to abstain from sperm donation from Day 1 through 90 days after the final dose of study drug;
   * Female patients of childbearing potential (ie, ovulating, pre-menopausal, and not surgically sterile) must have a documented negative serum pregnancy test at enrollment (Visit 1); and
   * Female patients of childbearing potential must use a highly effective method of contraception (ie, <1% failure rate) from Day 1 through 30 days after the last administration of study drug.
5. Are able and willing to give informed consent for participation in the clinical study.

Exclusion Criteria:

1. Have met Protocol-defined stopping criteria, were withdrawn from the study, discontinued CIN-107 at the time of Visits 6 or 9, or were not compliant with the Protocol during Study CIN-107-124;
2. Have received treatment with any investigational agent for disease intervention (ie, other than study drug) during Study CIN-107-124, or since the last administration of study drug in Study CIN-107-124, or plans to participate in another clinical study within 30 days of discontinuation of study drug;
3. Have had any new, significant, or uncontrolled comorbidity since initially enrolling in Study CIN-107-124 that would increase the risk of the patient in Study CIN-107-130, as determined by the Investigator;
4. Have had a mean seated SBP ≥170 mmHg or DBP ≥105 mmHg at the end of Part 1 or Part 2 of Study CIN-107-124;
5. Have an upper arm circumference that does not meet the cuff measurement criteria for the selected BP machine at Visit 1 of Study CIN-107-130;
6. Have any uncontrolled or clinically significant laboratory abnormality that would affect safety, interpretation of study data, or the patient's participation in the study, as determined by the Investigator;
7. Have experienced a de novo or reactivated serious viral infection such as hepatitis B, hepatitis C, or HIV during Study CIN-107-124;
8. Have had any major episode of infection requiring hospitalization or treatment with intravenous antibiotics during Study CIN-107-124;
9. Have developed a malignancy (with the exception of non-serious local and resectable basal or squamous cell carcinoma of the skin) during Study CIN-107-124;
10. Have anticipated initiation of erythropoietin-stimulating agents and/or planned transfusion within 2 months after enrollment (Visit 1);
11. Are expected to receive or are receiving any of the exclusionary drugs (strong cytochrome P450 3A inducers);
12. Have known secondary causes of HTN (eg, renal artery stenosis, uncontrolled or untreated hyperthyroidism, uncontrolled or untreated hypothyroidism, hyperparathyroidism, pheochromocytoma, Cushing's syndrome, or aortic coarctation) except obstructive sleep apnea;
13. Have been diagnosed with New York Heart Association stage III or IV chronic heart failure during Study CIN-107-124;
14. Have had a stroke, transient ischemic attack, hypertensive encephalopathy, acute coronary syndrome, or hospitalization for heart failure during Study CIN-107-124;
15. Have a known current severe left ventricular outflow obstruction, such as obstructive hypertrophic cardiomyopathy and/or severe aortic valvular disease diagnosed from a prior echocardiogram;
16. Have a planned coronary revascularization (percutaneous coronary intervention [PCI] or coronary artery bypass graft [CABG]) or any major surgical procedure;
17. Have had a CABG or other major cardiac surgery (eg, valve replacement), peripheral arterial bypass surgery, or PCI during Study CIN-107-124;
18. Have a planned dialysis or kidney transplant during the course of this study;
19. Have a known hypersensitivity to CIN-107 or drugs of the same class, or any of its excipients;
20. Have any clinically relevant medical or surgical conditions (including unstable conditions and/or treatment with systemic immunosuppressants including corticosteroids) that, in the opinion of the Investigator, would put the patient at risk by participating in the study;
21. Are pregnant, breastfeeding, or planning to become pregnant during the study; or
22. Are considered to be unsuitable for any other reason that may either place the patient at increased risk during participation or interfere with the interpretation of the study outcomes by the Investigator, after reviewing medical and psychiatric history, physical examination, and laboratory evaluation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Research Site, Saraland, Alabama
  - Research Site, Huntington Park, California
  - Research Site, Lincoln, California
  - Research Site, Los Angeles, California
  - Research Site, Northridge, California
  - Research Site, Oceanside, California
  - Research Site, Panorama City, California
  - Research Site, Van Nuys, California
  - Research Site, Clearwater, Florida
  - Research Site, Doral, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Miami, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Winter Haven, Florida
  - Research Site, Addison, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Morton, Illinois
  - Research Site, Brownsburg, Indiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Troy, Michigan
  - Research Site, Olive Branch, Mississippi
  - Research Site, Brooklyn, New York
  - Research Site, Columbus, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Austin, Texas
  - Research Site, Carrollton, Texas
  - Research Site, Dallas, Texas
  - Research Site, Georgetown, Texas
  - Research Site, Houston, Texas
  - Research Site, Lampasas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, West Valley City, Utah
  - Research Site, Manassas, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CIN-107-130&attachmentIdentifier=d0050f33-49b7-420e-85b3-72bc242fb2f8&fileName=CIN-107-130_StatisticalAnalysisPlan_redacted.pdf&versionIdentifier=
- See also: redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CIN-107-130&attachmentIdentifier=60503b71-c6c2-4618-a7da-9b419d900f40&fileName=CIN-107-130_CSP_redacted.pdf&versionIdentifier=
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CIN-107-130&attachmentIdentifier=0a211342-96b6-4917-8bb8-ec3489a54f7d&fileName=CIN-107-130_CSR_synopsis_redacted.pdf&versionIdentifier=
- Available data/document: Trial Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25790&tenant=MT_MED_9011 — Trial Results Summary

RESULTS

PARTICIPANT FLOW:
Groups:
- 2mg CIN-107: Participants received 2mg CIN-107 with potential of additional single background antihypertensive agent. Single background antihypertensive (non-CIN-107) agent chosen at Visit 1 or 2 should remain stable until Visit 3 of the study, after which the Investigator was permitted to use his/her medical judgment to up/down titrate or discontinue the background antihypertensive (non-CIN-107) agent.
Period: Overall Study
Arm/Group | 2mg CIN-107
Started | 175
Completed | 146
Not Completed | 29
Not completed — Lost to Follow-up | 6
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 19
Not completed — Noncompliance, Subject unable to complete last visit. | 3

BASELINE CHARACTERISTICS:
Arm/Group | 2mg CIN-107
Number analyzed (Participants) | 175
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The safety analysis set population
  Years | 60.6 (10.4)
Age, Customized [Number; unit: Participants] — Population: The safety analysis set population
  Participants
    > 75 years | 11
    <= 75 years | 164
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The safety analysis set population
  Participants
    Female | 78
    Male | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The safety analysis set population
  Participants
    Hispanic or Latino | 99
    Not Hispanic or Latino | 76
    Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Population: The safety analysis set population
  Participants
    American Indian or Alaska Native | 0
    Asian | 4
    Black or African American | 42
    Native Hawaiian or other Pacific Islander | 0
    Other | 1
    White | 128

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participants administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and/or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational medicinal product, whether or not related to the investigational medicinal product.
  Any medical condition already present at enrollment should be recorded as medical history and not be reported as an AE unless the medical condition or signs or symptoms present at baseline changes in severity, frequency, or seriousness at any time during the study. In this case, it was be reported as an AE.
Time Frame: 52 weeks
Population: Safety Population includes any participants enrolled in the study who have taken at least 1 dose of any study drug.
Measure: Number; unit: Participants
Arm/Group | 2mg CIN-107
Number analyzed (Participants) | 175
Participants | 73

2. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Events of Special Interest (AESIs)
Description: For this study, AESIs include the following:
  Events of hypotension that require clinical intervention; Abnormal potassium laboratory values that require clinical intervention; and Abnormal sodium laboratory values that require clinical intervention.
Time Frame: 52 weeks
Population: Safety Population includes any participants enrolled in the study who have taken at least 1 dose of any study drug.
Measure: Number; unit: Participants
Arm/Group | 2mg CIN-107
Number analyzed (Participants) | 175
Participants | 7

3. Primary Outcome: Number of Participants With Any Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was or adverse reaction is considered serious if, in the view of either the Investigator or Sponsor, it results in any of the following outcomes: Death, a life-threatening AE, a persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, a congenital anomaly/birth defect, or an important medical event.
Time Frame: 52 weeks
Population: Safety Population includes any participants enrolled in the study who have taken at least 1 dose of any study drug.
Measure: Number; unit: Participants
Arm/Group | 2mg CIN-107
Number analyzed (Participants) | 175
Participants | 8

4. Primary Outcome: Change From Baseline in Serum Potassium
Description: Mean change from baseline at Week 52 in serum potassium (mmol/L).
Time Frame: 52 weeks
Population: Safety Population includes any participants enrolled in the study who have taken at least 1 dose of any study drug. In the safety population 48 participants did not have baseline measure and/or 52 weeks measure for serum potassium.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 2mg CIN-107
Number analyzed (Participants) | 127
mmol/L | 0.08 (0.417)

5. Primary Outcome: Change From Baseline in Serum Sodium
Description: Mean change from baseline at Week 52 in serum sodium (mmol/L).
Time Frame: 52 weeks
Population: Safety Population includes any participants enrolled in the study who have taken at least 1 dose of any study drug. In the safety population 48 participants did not have baseline measure and/or 52 weeks measure for serum sodium.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 2mg CIN-107
Number analyzed (Participants) | 127
mmol/L | 0.6 (3.02)

6. Secondary Outcome: Change From Baseline in Mean Seated Systolic Blood Pressure
Description: Mean change from baseline at Week 52 in seated systolic blood pressure (SBP)
Time Frame: 52 weeks
Population: Safety Population includes any participants enrolled in the study who have taken at least 1 dose of any study drug. In the safety population 37 participants did not have 52 weeks measure for seated SBP.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 2mg CIN-107
Number analyzed (Participants) | 138
mmHg | -5.1 (11.51)

7. Secondary Outcome: Change From Baseline in Mean Seated Diastolic Blood Pressure
Description: Mean change from baseline at 52 weeks in mean seated diastolic blood pressure (DBP)
Time Frame: 52 weeks
Population: Safety Population includes any participants enrolled in the study who have taken at least 1 dose of any study drug. In the safety population 37 participants did not have 52 weeks measure for seated DBP.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 2mg CIN-107
Number analyzed (Participants) | 138
mmHg | -3.6 (8.65)

8. Primary Outcome: Change From Baseline in Body Weight
Description: Change from baseline at 52 weeks in body weight (kg)
Time Frame: 52 weeks
Population: Safety Population includes any participants enrolled in the study who have taken at least 1 dose of any study drug. In the safety population 37 participants did not have 52 weeks measure for body weight.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | 2mg CIN-107
Number analyzed (Participants) | 138
kg | -0.30 (3.839)

9. Primary Outcome: Change From Baseline in Temperature
Description: Change from baseline at 52 weeks in temperature (C)
Time Frame: 52 weeks
Population: Safety Population includes any participants enrolled in the study who have taken at least 1 dose of any study drug. In the safety population 37 participants did not have 52 weeks measure for temperature.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | 2mg CIN-107
Number analyzed (Participants) | 138
Celsius | -0.03 (0.473)

10. Primary Outcome: Change From Baseline in Seated Heart Rate
Description: Change from baseline at 52 weeks in seated heart rate (beats/min)
Time Frame: 52 weeks
Population: Safety Population includes any participants enrolled in the study who have taken at least 1 dose of any study drug. In the safety population 37 participants did not have 52 weeks measure for seated heart rate.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | 2mg CIN-107
Number analyzed (Participants) | 138
beats/min | 0.9 (9.49)

11. Secondary Outcome: Achieving Mean Seated Systolic Blood Pressure <130 mmHg
Description: Number of participants achieved mean seated systolic blood pressure (SBP) <130 mmHg at 52 week
Time Frame: 52 weeks
Population: Safety Population includes any participants enrolled in the study who have taken at least 1 dose of any study drug.
Measure: Number; unit: Participants
Arm/Group | 2mg CIN-107
Number analyzed (Participants) | 175
Participants | 102

12. Secondary Outcome: Non-responders in Study CIN-107-124 Achieving a Seated SBP Response <130 mmHg
Description: Number of non-responders (participants with seated SBP >=130 mmHg) in Study CIN-107-124 achieving a seated SBP response <130 mmHg with CIN-107 with/without a single background antihypertensive agent and/or rescue medication and irrespective of Study CIN-107-124 dose strength.
Time Frame: 52 weeks
Population: Subpopulation of the safety population (any participants enrolled in the study who have taken at least 1 dose of any study drug) who were non-responders (participants with seated SBP >=130 mmHg) in Study CIN-107-124.
Measure: Number; unit: Participants
Arm/Group | 2mg CIN-107
Number analyzed (Participants) | 53
Participants | 20

13. Secondary Outcome: Responders in Study CIN-107-124 Achieving a Seated SBP Response <130 mmHg
Description: Number of responders (participants with <130 mmHg) in Study CIN-107-124 achieving a seated SBP response <130 mmHg with CIN-107 with/without a single background antihypertensive agent and/or rescue medication and irrespective of Study CIN-107-124 dose strength.
Time Frame: 52 weeks
Population: Subpopulation of the safety population (any participants enrolled in the study who have taken at least 1 dose of any study drug) who were responders (participants with seated SBP <130 mmHg) in Study CIN-107-124.
Measure: Number; unit: Participants
Arm/Group | 2mg CIN-107
Number analyzed (Participants) | 122
Participants | 82

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | 2mg CIN-107
All-Cause Mortality (participants affected / at risk) | 0/175
Serious Adverse Events (participants affected / at risk) | 8/175
Other Adverse Events (participants affected / at risk) | 20/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2mg CIN-107 (N=175)
Lacunar stroke (Nervous system disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Femoral nerve injury (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2mg CIN-107 (N=175)
Urinary tract infection (Infections and infestations) | 13 (16)
Hyperkalaemia (Metabolism and nutrition disorders) | 9 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less or equal to 60 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication and can extend the embargo for up to 90 days.

DOCUMENTS (2):
  • Study Protocol (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/88/NCT05459688/Prot_002.pdf
  • Statistical Analysis Plan (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT05459688/SAP_003.pdf